CLINICAL TRIAL: NCT00881322
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Parallel-Group Clinical Trial to Evaluate the Effects of Gas Defense On Intestinal Gas Symptoms in Otherwise Healthy Adults
Brief Title: A Study on Intestinal Gas Symptoms to Evaluate the Effects of Gas Defense in Otherwise Healthy Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami Research Associates (Network)
Collaborators: Ganeden Biotech, Inc. (Industry)
Responsible Party: Diane Krieger, MD - Principal Investigator, Miami Research Associates
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GAN-2008
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Abdominal Pain; Abdominal Cramps; Flatulence
MeSH Terms: conditions — Abdominal Pain; Colic; Flatulence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BC-130 (Experimental): Active Arm
  Interventions: Dietary Supplement: BC-130 (Gas Defense)
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BC-130 (Gas Defense) — Product Dosing:
  Take one capsule daily, at approximately the same time of day, without regard to food (may be taken with or without food)
  Gas Defense Serving Size: 1 tablet Active Ingredients: B. Coagulans, Enzyme Blend (Cellulase - Trichoderma longibrachiatum, Cellulase - Aspergillus niger, Hemicellulase, Alpha Galactosidase, Invertase) Inactive Ingredients: vegetable capsule, Magnesium Stearate, Silicon Dioxide, Maltodextrin Contains: Wheat, Fish.
  Other Names: Gas Defense
  Arms: BC-130
Dietary Supplement: Placebo — Product Dosing:
  Take one capsule daily, at approximately the same time of day, without regard to food (may be taken with or without food)
  Placebo - matched in size and color to the active product Inactive Ingredients: microcrystalline cellulose, FD&C yellow #5 Lake, FD&C blue #1 Lake, FD&C red #46 Lake and vegetable capsule
  Arms: Sugar Pill

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to determine the safety and efficacy of Digestive Advantage™ Gas Defense formula, a probiotic dietary supplement. The study will last approximately four weeks, and subjects will be seen at a screening/randomization visit, and two follow-up visits.

Study procedures will include administering questionnaires for assessment of the study product's effect on intestinal gas symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-75 years of age.
* Subject self-reports at least one of the following symptoms after eating a meal or snack:
* Abdominal pain/cramps
* Distended feeling/bloating
* Flatulence/gas
* Subject is in otherwise general good health as determined by physical exam and medical history.
* Subject is willing and able to comply with the protocol.
* Female subjects not defined as post-menopausal (excluding hysterectomized and post bilateral tubal ligations) must use a reliable method of birth control as defined within this protocol.
* Subject is able to understand and sign the informed consent (English or Spanish) to participate in the study.

Exclusion Criteria:

* Subject has any of the following medical conditions:

  * active heart disease
  * renal or hepatic impairment/disease
  * Type I or II diabetes
  * psychiatric disorders (hospitalized within the past one year)
  * bipolar disorder
  * Parkinson's disease
  * unstable thyroid disease
  * immune disorder (such as HIV/AIDS)
  * any medical condition deemed exclusionary by the Principal Investigator (PI)
* Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within five years prior to screening.
* Subject has had any stomach or intestinal surgery (i.e. gastric bypass).
* Subject is currently taking antibiotics (or any drug that significantly interferes with bacterial flora) or has taken antibiotics within the 30 days prior to screening/enrollment.
* Subject is currently taking or has used in the past 30 days probiotics or prebiotics.
* Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).
* Subject is currently taking any medication deemed exclusionary by PI.
* Subject has a history of or currently has any gastrointestinal disorders or inflammatory bowel conditions such as Crohn's disease, short bowel, or ulcerative colitis. Subjects may not have a diagnosis, be seeing a doctor, or taking prescription medication(s) for Irritable Bowel Syndrome (IBS).
* Subject has constipation defined as less than three spontaneous bowel movements per week.
* Subject is lactose intolerant (self-professed or diagnosed).
* Subject uses any of the following classification of GI medications two or more times per week: anti-spasmodics, motility agents, pro-kinetic agents or laxatives.
* Subject plans to use another over-the-counter gas-relief product daily during the study period. Over-the-counter gas relief products may be used as rescue medication (their use will be captured by the study staff). If a subject is using a fiber supplement prior to starting the study, he/she may continue as long as the frequency and quantity remain stable throughout the study period.
* Subject has an allergy to wheat or fish or any of the other product ingredients (see section 2.5.4).
* Subject has two or more food allergies.
* Subject has a history of drug or alcohol abuse within the past 12 months.
* Subject is deemed by the Investigator as an unsuitable candidate for receipt of an investigational dietary supplement, or unable to be followed up throughout the entire duration of the study.
* Female subject of childbearing potential is unwilling to use an acceptable form of contraceptive device throughout the study period.
* Subject is pregnant, lactating, or planning to become pregnant during the study period.
* Subject is participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment.
* Subject is deemed by the Investigator as an unsuitable candidate for receipt of an investigational dietary supplement, or unable to be followed up throughout the entire duration of the study.
* Subject is unable to comprehend the Informed Consent and research purpose.
* Subject is unable or unwilling to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of daily supplementation with GD as compared to placebo on intestinal gas symptoms as measured by the subscores of the GI Symptom Rating Scale (GSRS) and the subscores of the Severity of Dyspepsia Assessment (SODA). | 4 weeks
Primary Safety Objective To determine if daily supplementation with GD is safe within the confines of this study as denoted by changes from baseline in blood pressure, heart rate, adverse events, and subjective remarks. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane Krieger, MD, Principal Investigator — Medical Director
Locations (2):
- Miami Research Associates, Miami, Florida, United States
- Latin American Research, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Kalman DS, Schwartz HI, Alvarez P, Feldman S, Pezzullo JC, Krieger DR. A prospective, randomized, double-blind, placebo-controlled parallel-group dual site trial to evaluate the effects of a Bacillus coagulans-based product on functional intestinal gas symptoms. BMC Gastroenterol. 2009 Nov 18;9:85. doi: 10.1186/1471-230X-9-85. PMID 19922649